CLINICAL TRIAL: NCT05044390
Title: Lung Transplantation for Pleuroparenchymal Fibroelastosis : a French Multicentric Retrospective Study
Brief Title: Lung Transplantation for Pleuroparenchymal Fibroelastosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 420
Record Dates: First submitted 2021-08-30; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Fibroelastosis
MeSH Terms: interventions — Lung Transplantation; Single Person

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung transplantation: Lung transplantation performed for end-stage interstitial lung disease secondary to pleuroparenchymal fibroelastosis.
  Interventions: Procedure: Lung transplantation (single, lobar or bilateral lung transplantation)

INTERVENTIONS:
Procedure: Lung transplantation (single, lobar or bilateral lung transplantation) — Lung transplantation were performed for end-stage interstitial lung disease secondary to pleuroparenchymal fibroelastosis

SUMMARY:
This retrospective observational study will evaluate the outcomes of lung transplantation for a rare cause of interstitial lung disease called pleuroparenchymal fibroelastosis. Data will be collected from all transplantation center in France.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplantation (any type) for pleuroparenchymal fibroelastosis
* Histologically confirmed pleuroparenchymal fibroelastosis on the recipient lungs

Exclusion Criteria:

* All other interstitial lung disease than pleuroparenchymal fibroelastosis
* Pleuroparenchymal fibroelastosis who didn't underwent lung transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pleuroparenchymal fibroelastosis who underwent lung transplantation in France between 2005 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative mortality | Any death up to 90 days after lung transplantation
  Any death after lung transplantation during the first 30 days or during the hospitalization following the lung transplantation (in-hospital mortality)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Marie Lannelongue Hospital, Le Plessis-Robinson
  - Hopital Louis Pradel, Lyon
  - Bichat Claude Bernard Hospital, APHP, Paris
  - Foch Hospital, Suresnes

REFERENCES:
- [Derived] Clermidy H, Mercier O, Brioude G, Mordant P, Fadel G, Picard C, Chatron E, Le Pavec J, Roux A, Reynaud-Gaubert M, Messika J, Olland A, Demant X, Degot T, Lavrut PM, Jougon J, Sage E, Fadel E, Thomas P, Cottin V, Tronc F. Outcomes of lung transplantation for pleuroparenchymal fibroelastosis: A French multicentric retrospective study. J Heart Lung Transplant. 2024 Oct;43(10):1727-1736. doi: 10.1016/j.healun.2024.06.009. Epub 2024 Jun 21. PMID 38909712